CLINICAL TRIAL: NCT00087776
Title: Phase III Study of Taxoprexin Injection vs. Dacarbazine in Patients With Metastatic Malignant Melanoma
Brief Title: Study of Taxoprexin Injection vs. Dacarbazine in Patients With Metastatic Malignant Melanoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis determined that the futility boundary had been crossed and there was no reasonable prospect that statistical significance would be achieved if patient accrual continued
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01-02-17
Record Dates: First submitted 2004-07-13; First posted 2004-07-16 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2018-01

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — docosahexaenoyl-paclitaxel; Docosahexaenoic Acids; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Taxoprexin (Experimental): Taxoprexin® 900 mg/m² intravenously every 3 weeks
  Interventions: Drug: Taxoprexin
- Dacarbazine (Active Comparator): Dacarbazine 1000 mg/m² intravenously every 3 weeks.
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: Taxoprexin — Administered by intravenous infusion over 2 hour infusion on Day 1 followed by a 20-day observation period for a total of 21 days (three weeks) per course
  Other Names: Docosahexaenoic acid (DHA)-paclitaxel
  Arms: Taxoprexin
Drug: Dacarbazine — Administered by intravenous infusion over 30 minutes on Day 1 followed by a 20-day observation period for a total of 21 days (three weeks) per course
  Other Names: Imidazole carboxamide
  Arms: Dacarbazine

SUMMARY:
The primary objective of this trial is to compare the survival of patients with metastatic malignant melanoma treated with Taxoprexin Injection to those treated with Dacarbazine. In addition, the response rate to each drug, response duration, time to progression and time to treatment failure will be measured. Toxicity will be evaluated and compared between the two groups.

DETAILED DESCRIPTION:
This was a randomized, multi-center, open-label Phase III study in patients with histologically confirmed metastatic malignant melanoma. Patients received either Taxoprexin® at a starting dose of 900 mg/m2 intravenously by 2-hour infusion on Day 1 every 3 weeks or dacarbazine at a starting dose of 1000 mg/m2 intravenously over at least 30 minutes once every 3 weeks. Treatment continued until progression of disease, intolerable toxicity, refusal of continued treatment by the patient, or, in the investigator's opinion, treatment discontinued. Disease status was assessed every 6 to 8 weeks using standard imaging techniques. All images were forwarded to the sponsor and archived. Following the end of protocol treatment, further treatment was at the investigator's discretion but no cross-over was planned. All patients were followed until death

ELIGIBILITY:
Inclusion Criteria:

* Patients must have malignant melanoma, and documented metastatic disease.
* Patients must have at least one unidimensionally measurable lesion.
* Patients must not have received prior systemic chemotherapy for metastatic disease. Prior treatment with immunotherapy or vaccine therapy is allowed provided there is documentation of disease progression.
* At least 6 weeks (42 days) since any prior immunotherapy, cytokine, biologic, vaccine or other therapy unless patients have progressed during immunotherapy.
* At least 4 weeks (28 days) since any prior radiotherapy.
* Lesions being used to assess disease status may not have been radiated.
* Patients must have Eastern Cooperative Oncology Group performance status of 0 - 2.
* Patients must be >= 18 years of age.
* Patients must have adequate renal and liver function
* Patients must have adequate bone marrow function.
* Life expectancy of at least 3 months.
* Patients must sign an informed consent form indicating that they are aware of the investigational nature of this study and in keeping with the policies of the institution.

Exclusion Criteria:

* Patients who have received prior therapy with any taxane or dacarbazine.
* Patients whose primary site is the eye.
* Patients who have a past or current history of neoplasm other than the entry diagnosis, except for curatively treated non-melanoma skin cancer or carcinoma in situ of the cervix or other cancers cured by surgery alone with a disease-free survival longer than 5 years.
* Patients with uncontrolled brain metastasis.
* Patients who are pregnant or nursing and patients who are not practicing an acceptable method of birth control. Patients may not breastfeed while on this study.
* Patients with current active infections requiring anti-infectious treatment (e.g., antibiotics, antivirals, or antifungals).
* Patients with current peripheral neuropathy of any etiology that is greater than grade 1.
* Patients with unstable or serious concurrent medical conditions are excluded.
* Patients with a known hypersensitivity to Cremophor.
* Patients must not have had recent major surgery within the past 14 days or large field radiation therapy, chemotherapy, endocrine therapy in the last 28 days, or biologic therapy in the last 42 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2002-12-06 (Actual); Primary Completion 2007-10-27 (Actual); Study Completion 2007-10-27 (Actual)

PRIMARY OUTCOMES:
Overall Participant Survival | Up to 36 months
  Overall survival was defined as the time from the day of randomization to participant death or the termination of the study, whichever occurs first. Participants were contacted monthly for survival information.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieved an Objective Complete Response or Partial Response | Assessed every 6 weeks, up to 38 months
  Antitumor response was defined as the percentage of participants who achieved an objective response (Confirmed Response [CR] or Partial Response [PR]), confirmed by repeat assessments performed no less than 4 weeks after the criteria for response were first met. Response was based on the blinded radiological review using Response Evaluation Criteria in Solid Tumors (RECIST) response guidelines, Version 1.0. A complete response was defined as a disappearance of all target lesions determined by 2 consecutive observations not less than 4 weeks apart. Partial response was defined as a 30% decrease in the sum of the longest diameters (LD) of target lesions, taking as reference the baseline sum of LD determined by 2 consecutive observations not less than 4 weeks apart.
Duration of Response | Assessed every 6 weeks, up to 36 months
  Duration of overall response was a measurement from the time measure criteria was met for confirmed complete response or partial response (whichever was first recorded) until the first date that recurrent of progressive disease was objectively documented (taking as reference for progressive disease the smallest measurement recorded since treatment started).
Time to Progression (TPP) | Assessed every 6 weeks until progression or death, up to 36 months
  Progression free survival time was defined as the time from the day of randomization to the start of documented progression, based on the blinded radiological review response assessment. Progressive disease was defined as a ≥ 20% increase in the sum of longest diameter (SLD) of target lesions, taking as reference the smallest SLD recorded since the treatment started or the appearance of one or more new lesions
Time to Failure (TTF) | Baseline to stopping treatment, up to 36 months
  Time to Failure (TTF) was defined as the time from the day of randomization to the discontinuation of protocol treatment for any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals, Inc., Norristown, Pennsylvania, United States